CLINICAL TRIAL: NCT01575535
Title: S0106B, Stem Cell Origin in AML: Prognostic and Therapeutic Implications
Brief Title: S0106B Studying Bone Marrow Samples From Women With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: S0106B; S0106B (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2012-04-10; First posted 2012-04-11 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Leukemia
Keywords: untreated adult acute myeloid leukemia; adult acute basophilic leukemia; adult acute eosinophilic leukemia; adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute megakaryoblastic leukemia (M7); adult acute minimally differentiated myeloid leukemia (M0); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with del(5q); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myelomonocytic leukemia (M4)
MeSH Terms: conditions — Leukemia; Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute | interventions — Gene Expression Profiling; Flow Cytometry

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: gene expression analysis
Other: flow cytometry
Other: fluorescence activated cell sorting
Other: laboratory biomarker analysis
Other: medical chart review

SUMMARY:
RATIONALE: Studying samples of bone marrow from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer.

PURPOSE: This research trial studies bone marrow samples from women with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Estimate the proportion of acute myeloid leukemia (AMLs) that originate in CD33+ precursors or in which uncontrolled growth is limited to CD33+ precursors.
* Explore whether there is an association between the cellular origin of AML (i.e., origination in CD33+ precursors or not) and cytogenetic, molecular, and other patient characteristics.
* Explore whether overall survival (OS), event-free survival (EFS), disease-free survival (DFS), response rate (RR), or relapse rate is improved for patients with AMLs that originate in CD33+ precursors or in which uncontrolled growth is limited to CD33+ precursors compared to patients with clonally involved cells not detected.

OUTLINE: Archived bone marrow samples are analyzed for CD33+ progenitors, X-chromosome inactivation, and somatic mutations (t(8;21), inv(16), FLT3/ITD, NPM1, CEBPA, KIT) by fluorescence-activated cell sorting, long-term culture in hypoxic condition in cytokine-containing liquid media, and flow cytometry. Results are then compared with each patient clinical data.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnostic bone marrow specimens from female patients with untreated AML undergoing intensive ("3+7"-like) induction chemotherapy
* Specimens from the South Western Oncology Group (SWOG) protocols S0106 (age 18 to 60 years), excluding patients who received gemtuzumab ozogamicin (GO), and S9333 (age > 60 years)

PATIENT CHARACTERISTICS:

* See Disease Characteristics

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Repository specimens
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Association between CD33+ precursors and cytogenetic and/or molecular risks using Fisher's exact test | May 2012
Relationship between emergence of individual mutations [t(8;21), inv(16), FLT3/ITD, NPM1, CEBPA, and KIT], clonality, and stage of cell differentiation using Fisher's exact test | May 2012
Associations between survival outcomes (OS, EFS, DFS, RR, and relapse rate) and CD33+ restriction using regression analysis | May 2012

CONTACTS AND LOCATIONS:
Overall Officials: Roland Walter, MD, PhD, Principal Investigator — Fred Hutchinson Cancer Center